CLINICAL TRIAL: NCT01868126
Title: A Phase II, Randomized, Observer-masked, Placebo-and Active-controlled, Parallel-group, Multi-center Study Assessing the Safety and Efficacy of DE-117 Ophthalmic Solution Compared With Latanoprost and Placebo in Subjects With Primary Open-angle Glaucoma or Ocular Hypertension
Brief Title: Multi-center Study Assessing the Safety and Efficacy of DE-117 Ophthalmic Solution in Subjects With Primary Open-angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Santen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 33-002
Record Dates: First submitted 2013-05-29; First posted 2013-06-04 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Open-angle Glaucoma or Ocular Hypertension
Keywords: Santen; Eye; Glaucoma; Ocular hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group 1: DE-117 ophthalmic solution (Experimental): One drop DE-117 Low Dose in each eye daily for 28 days
  Interventions: Drug: DE-117 ophthalmic solution
- Group 2: DE-117 ophthalmic solution (Experimental): One drop DE-117 Low Middle Dose in each eye daily for 28 days
  Interventions: Drug: DE-117 ophthalmic solution
- Group 3: DE-117 ophthalmic solution (Experimental): One drop DE-117 High Middle Dose in each eye daily for 28 days
  Interventions: Drug: DE-117 ophthalmic solution
- Group 4: DE-117 ophthalmic solution (Experimental): One drop DE-117 High Dose in each eye daily for 28 days
  Interventions: Drug: DE-117 ophthalmic solution
- latanoprost ophthalmic solution (Active Comparator): One drop latanoprost 0.005% in each eye daily for 28 days
  Interventions: Drug: latanoprost ophthalmic solution
- placebo (vehicle of DE-117) ophthalmic solution (Placebo Comparator): One drop DE-117 vehicle in each eye once daily for 28 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: DE-117 ophthalmic solution
  Arms: Group 1: DE-117 ophthalmic solution; Group 2: DE-117 ophthalmic solution; Group 3: DE-117 ophthalmic solution; Group 4: DE-117 ophthalmic solution
Drug: latanoprost ophthalmic solution
  Arms: latanoprost ophthalmic solution
Other: Placebo
  Arms: placebo (vehicle of DE-117) ophthalmic solution

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of four concentrations of DE-117 ophthalmic solution.

DETAILED DESCRIPTION:
This is a 28-day randomized, observer-masked, placebo-and active-controlled, parallel-group, multi-center, study investigating the safety and efficacy of four concentrations of DE-117 ophthalmic solution when compared to latanoprost (0.005% latanoprost) and placebo (vehicle of DE-117) in subjects with primary open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Main Inclusion Criteria:

* Current diagnosis of primary open-angle glaucoma or ocular hypertension in both eyes
* Qualifying intraocular pressure in at least one eye at Baseline
* Qualifying corrected ETDRS visual acuity in each eye
* Qualifying central cornea thickness in each eye

Main Exclusion Criteria:

* Closed/barely open anterior chamber angle or a history of acute angle closure in either eye
* Diagnosis of primary open-angle glaucoma or ocular hypertension due to etiology known to be non-responsive to conventional drug therapy
* Evidence of advanced glaucoma, visual field defect or progressive visual field loss that that do not meet the study criteria
* History of ocular surgery specifically intended to lower IOP
* History of any ocular or systemic abnormality or condition that may put the subject at significant risk, may confound study results, or may interfere significantly with the subject's participation in the study
* Intended or current use of any ocular medications other than study medications during the study
* Use of contact lenses within one week prior to Baseline (Day 1) until end of treatment
* Known allergy or sensitivity to any components of the study medications
* Use of steroids (systemic) within 30 days prior to Visit 1 (Screening)
* Anticipate the need to initiate or modify an existing chronic therapy that could substantially affect IOP or the study outcomes during the study period
* Females who are pregnant, nursing or planning a pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2013-05; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure (mmHg) | Day 1, Day 8, Day 15 and Day 29
  Intraocular pressure (mmHg) measurements will be collected at each visit using Goldmann applanation tonometry

SECONDARY OUTCOMES:
Adverse events | Day 1, Day 8, Day 15 and Day 29
  Adverse events will be assessed at each visit to evaluate safety
Ocular signs and symptoms | Day 1, Day 8, Day 15 and Day 29
  Ocular symptoms and ocular signs will be collected at each visit using slit lamp biomicroscopy, dilated ophthalmoscopy, gonioscopy, automated perimetry visual field testing, corrected visual acuity and pachymetry

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Newport Beach, California
  - Morrow, Georgia
  - Kansas City, Missouri
  - Rochester, New York
  - Cleveland, Ohio
  - Austin, Texas
  - San Antonio, Texas